CLINICAL TRIAL: NCT04775004
Title: Comparing Meniscal Repair Biologic Augmentation: Marrow Venting Procedure Versus PRP (MVP Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: American Orthopaedic Society for Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB20-1394
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Meniscal Tear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone marrow venting procedure (BMVP) (Active Comparator): Subjects randomized in the OR to undergo BMVP surgical augmentation
  Interventions: Other: Bone marrow venting procedure (BMVP)
- Platelet rich plasma (PRP) (Active Comparator): Subjects randomized in the OR to undergo PRP surgical augmentation
  Interventions: Other: Platelet Rich Plasma (PRP)

INTERVENTIONS:
Other: Bone marrow venting procedure (BMVP) — The BMVP involves creating small holes in a non-weight bearing area of the bone that does not have any important structures; the holes act as channels, which allow for flow of the participants own biologic products and stem cells from within the bone marrow.
  Arms: Bone marrow venting procedure (BMVP)
Other: Platelet Rich Plasma (PRP) — The PRP group will have 40cc to 60cc (about 3 tablespoons) of blood drawn at the time of surgery. The blood sample will then be prepared in a centrifuge machine to collect a component of the blood called platelet rich plasma. Once appropriate concentrations of the PRP are confirmed, the PRP will be injected into the subject's knee prior to wound closure.
  Arms: Platelet rich plasma (PRP)

SUMMARY:
There are no current or past RCT comparing biologic augments for meniscal repair. There is good data supporting both the use of BMVP of the intercondylar notch and intra-articular PRP injections for augmentation of meniscal repair. However, the effectiveness of these augmentation methods with respect to each other has never been investigated. The knowledge gained will allow us to potentially influence and adapt protocols to treat this particular patient population. Additionally, resources available at our institution provide a supportive framework with which to maintain contact with patients after hospital discharge. These key factors will allow us to perform a robust analysis of this population, to include outcomes measures of function as well as meniscal repair failure and reoperation rate.

The proposed interventional aim to compare meniscal repair augmentation methods is novel, as the direct comparison of these outcome measures has not been previously described. Because of the known benefit of biologic augmentation of meniscal repair, the investigators hypothesize that the repair failure rate for both cohorts will be lower than the reported repair failure rate for isolated tears without biologic augmentation; the investigators also hypothesize that BMVP of the intercondylar notch will clinically be significantly better than intra-articular PRP injection. The basis behind this hypothesis is in vivo evidence as well as a small RCT supporting the use of BMVP as augmentation for meniscal repair procedures.

ELIGIBILITY:
Inclusion Criteria

1. Age 16 or older
2. Medial, lateral, vertical longitudinal, oblique, or radial meniscal tear
3. Complex tears may be included at the discretion of the site investigator if patient has one of tear patterns listed in inclusion criteria 2 as the most predominant finding
4. No other concomitant procedure unless one of the following:

   * Chondroplasty
   * Synovectomy
   * Loose body removal
   * "Contralateral" menisectomy (i.e. medial meniscus repair with a lateral menisectomy or lateral meniscus repair with a medial menisectomy) would be permitted for inclusion
   * Any other procedure that does not include drilling, requires prior approval of the study sponsor for each procedure

Exclusion Criteria

1. Patients requiring cartilage restorative or repair procedures (i.e. OCD fixation, micro-fracture repair, or others)
2. Patients with meniscus root tears
3. Patients undergoing repair for horizontal cleavage tears
4. Kellgren-Lawrence scale 3>
5. Patients undergoing lateral release
6. Ipsilateral chondral lesion with Outerbridge classification of 3-4
7. Use of prednisone or other steroids, any immunosuppressant, or chemotherapy 1-week before surgery or expected use within six weeks after surgery
8. Cortisone use within the six weeks prior to surgery
9. Utilizing worker's compensation at the time of screening
10. Any previous ligament surgery on the index limb. Any previous meniscal surgery on the index meniscus.
11. Concomitant ligamentous insufficiency
12. Inflammatory rheumatic disease or other rheumatic disease
13. Immune compromised patients (hepatitis, HIV, etc.)
14. Any nicotine based products within the three months prior to surgery (including cigarettes, cigars, vaping, nicotaine patch, etc)
15. History of distal femur, proximal tibia, or patellar fracture that was treated operatively
16. Non English-speaking patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Promis Physical function CAT lower extremity score | 1-year after meniscus tear operation.
  Adaptive questionnaire that takes five minutes or less to complete and helps record how subject injury and recovery from surgery is affecting their normal life.

SECONDARY OUTCOMES:
Re-tear of repair meniscus | 1-year after meniscus tear operation.
  Clinically reported (symptomatic) and MRI confirmed via observation of fluid filled tear in the repaired tissue

CONTACTS AND LOCATIONS:
Overall Officials: Aravind Athiviraham, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.